CLINICAL TRIAL: NCT07304336
Title: Comparing the Efficacy of Dietary Strategies in Managing Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD): a Randomized Controlled Trial
Brief Title: Dietary Strategies for MASLD (Metabolic Dysfunction-Associated Steatotic Liver Disease)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, Associate Professor, MD, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MASLD_DIET
Record Dates: First submitted 2025-10-02; First posted 2025-12-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: MASLD
Keywords: Hepatic disorders; MASLD; Nutrition intervention
MeSH Terms: conditions — Digestive System Diseases | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Carb Diet (LCHO) (Experimental)
  Interventions: Behavioral: Low-Carb diet
- Mediterranean Diet (MeD) (Experimental)
  Interventions: Behavioral: Mediterranean diet
- Control group (Placebo Comparator)
  Interventions: Behavioral: Standard Lifestyle Recommendations

INTERVENTIONS:
Behavioral: Low-Carb diet — Participants followed a low-carbohydrate diet for 6 months. Macronutrient distribution: 35-40% carbohydrates, 30% protein, 30-35% fats. The diet was tailored based on participants' energy requirements.
  Arms: Low-Carb Diet (LCHO)
Behavioral: Mediterranean diet — Participants followed a Mediterranean-style diet for 6 months, providing 50-60% of energy from carbohydrates, approximately 15% from protein, and 25-35% from fat. The diet was tailored to individual energy requirements and patients in this group, should consume moderate portions of fish, poultry, and dairy products. The recommended cereal servings were larger than those for the LCHO arm.
  Arms: Mediterranean Diet (MeD)
Behavioral: Standard Lifestyle Recommendations — Participants received standard nutritional raccomandations for 6 months, including guidance on healthy eating, advices for regular physical activity, and educational materials consistent with standard clinical practice. No specific dietary plan was prescribed.
  Arms: Control group

SUMMARY:
This is a non-blinded, three-arm, parallel, 6-month randomized, longitudinal, and controlled intervention trial. designed to compare the effects of three dietary regimes (Mediterranean diet, low-carbohydrate diet and standard nutritional recommendations) on non-invasive parameters of fat accumulation and liver damage, including radiological and biochemical tests, in overweight or obese subjects with MASLD. Participants were enrollment and screening from the Liver Unit of the Department of Medical Sciences, University of Torino and randomly assigned to one of three groups: a low-carbohydrate diet, a mediterranean diet, or standard nutritional recommendations.

All participants were submitted to the following assessments both at enrollment and at after 6 month at the end of the study: 3-day food record; the Medi-Lite score; anthropometric measurements (weight, height, BMI, waist and neck circumferences); fat mass, fat-free mass by bioelectrical impedance; hand-grip strength; energy expenditure by indirect calorimetry; blood pressure measurement; blood sampling for metabolic variables and biomarkers of liver damage and liver disease measures (Cap, Stiffness and Fib-4).

DETAILED DESCRIPTION:
This is a three-arm, parallel-group, open-label randomized controlled trial designed to evaluate the effectiveness of three different nutritional interventions on non-invasive markers of liver damage, including radiological and biochemical assessments. Patients with MASLD were recruited from the Liver Unit of the Department of Medical Sciences, University of Torino.

At baseline, participants were randomly assigned to one of the following three groups:

A) Low-carb Diet (LCHO: 35-40% carbohydrates, 30% protein, 30-35% fats.) B) Mediterranean Diet (MeD: 50-60% carbohydrates, 15% protein, 25-35% fats ) C) Control group: standard nutritional recommendations The following evaluations were performed both at baseline and after 6 months at the and of the study: 3-day food record; the Medi-Lite score; anthropometric measurements (weight, height, BMI, waist and neck circumferences, fat mass, fat-free mass by bioelectrical impedance); hand-grip strength; energy expenditure by indirect calorimetry; blood pressure measurement; blood sampling for metabolic variables and biomarkers of liver damage and liver disease measures (Cap, Stiffness and Fib-4).

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 and <75 years
* BMI ≥25 and <35 kg/m2
* not having previously received nutritional advice for the liver disease

Exclusion Criteria:

* other causes of liver disease (including viral, autoimmune, cholestatic, genetic, alcoholic, and drug-induced)
* other diseases or conditions requiring specific dietary recommendations
* a history of alcohol abuse
* diabetes mellitus
* pharmacological treatments potentially interfering with study outcomes (corticosteroids, glucagon-like-peptide 1 agonists, biologic drugs)
* pregnancy or breastfeeding
* inability to give written informed consent
* life expectancy expected to be <1 year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Within- and between-group changes in hepatic steatosis [percentage, %] | 6 months
  The unit of measure is the percentage (%) of liver fat content, as assessed by transient elastography - FibroScan®.
Within- and between-group changes in Controlled Attenuation Parameter. (CAP) [dB/m] | 6 months
  The unit of measure is decibels per meter (dB/m), as measured by transient elastography - FibroScan®.

SECONDARY OUTCOMES:
Change in liver stiffness measured by transient elastography - FibroScan®. [kilopascals, kPa] | 6 months
  Liver stiffness will be assessed using transient elastography - FibroScan®.
Changes in fibrosis-4 index | 6 months
  Within- and between-group changes in fibrosis-4 index, a non-invasive score for liver fibrosis calculated by the following formula:
  FIB-4= (age x AST / (platelet count (x 10 9 ) x√ALT). This index has no fixed upper limit; higher values indicate worse fibrosis.
Changes in fat mass percentage | 6 months
  Within- and between-groups changes in fat mass percentage measured by bioelectrical impedance analysis
Changes in energy expenditure. | 6 months
  Within- and between-group changes in energy expenditure measured by indirect calorimetry.
Changes in insulin restistance [mmol/LxμU/mL] | 6 months
  Within- and between-group changes in HOMA-IR [mmol/LxμU/mL]
Changes in serum transaminase levels | 6 months
  Within- and between-group changes in serum transaminase levels [U/L]
Changes in thrombospondin-2 (TSP2) [ng/ml] | 6 months
  Assessing serum Thrombospondin-2 (TSP2) changes across incremental delta of weight loss
Changes in C-terminal procollagen 4 (PRO-C4) [ng/ml] | 6 months
  Assessing serum C-terminal procollagen 4 (PRO-C4) changes across incremental delta of weight loss

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino, University of Torino, Torino., Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT07304336/ICF_000.pdf